CLINICAL TRIAL: NCT00403325
Title: Phase I Study of Intravitreally Administered Ranibizumab in Subjects With Unresolving CSC and Subfoveal Fluid.
Brief Title: Intravitreal Ranibizumab Treatment of Central Serous Chorioretinopathy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vitreous -Retina- Macula Consultants of New York (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Richard Spaide, MD / Principal Investigator, Vitreous Retina Macula Consultants of New York
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FVF3850S
Record Dates: First submitted 2006-11-22; First posted 2006-11-23 (Estimated); Last update posted 2008-11-03 (Estimated); Status verified 2008-10

CONDITIONS: Central Serous Chorioretinopathy
Keywords: Central Serous Chorioretinopathy
MeSH Terms: conditions — Central Serous Chorioretinopathy | interventions — Ranibizumab

INTERVENTIONS:
Drug: rhuFab V2 [ranibizumab] ( Lucentis )

SUMMARY:
The purpose of this study is to examine the effects of Lucentis for active Central Serous Chorioretinopathy.

DETAILED DESCRIPTION:
This is an open-label, Phase I study of intravitreally administered ranibizumab in subjects with unresolving CSC and subfoveal fluid. Patients will be evaluated at baseline with ophthalmic examination, fluorescein angiography, optical coherence tomography, and color photography. Subjects will receive open-label intravitreal injections of 0.5 mg ranibizumab administered every 28 days (± 2 days) for 3 injections. Thereafter they are to be evaluated every month until month 12. Treatment will be administered to patients if there is presence of active leakage as determined by fluorescein angiography or persistence presence of sub retinal fluid upon OCT examination at that monthly visit.

ELIGIBILITY:
Inclusion Criteria:

* A history of persistent central serous chorioretinopathy present for at least 3 months Best-corrected visual acuity (BCVA) of 20/40 (73 letters on the ETDRS chart) to light perception as measured by ETDRS protocol refraction.
* No signs of choroidal neovascularization
* Documented subfoveal fluid by OCT
* Active leak associated with the subfoveal fluid
* The ability and willingness to provide written informed consent

Exclusion Criteria:

* Prior treatment with laser or PDT
* Have uncontrolled hypertension
* Have a history of thromboembolic events including stroke, transient ischemic attacks, and myocardial infarction
* Have use of or need for continued anticoagulation therapy, except aspirin 325 mg/day.
* Are receiving or require chronic concomitant therapy with systemic (> 5 mg) or topical ocular corticosteroids. Chronic concomitant therapy is defined as multiple doses taken daily for 14 or more consecutive days at any time within 6 months prior to screening
* Previously vitrectomized eyes.
* Had allergic reactions to fluorescein dye or lack of venous access.
* Any other additional ocular diseases which could irreversibly compromise the visual acuity of the study eye including amblyopia, anterior ischemic optic neuropathy (AION), age related macular degeneration (AMD), retinal detachment, severe cataracts, etc.
* An anticipated need for ocular surgery during the duration of the trial.
* Within 1 month prior to screening, have had intra ocular surgeries (including cataract surgery) in the study eye.
* Intravitreal triamcinolone or bevacizumab in the previous 2 months
* Uncontrolled glaucoma (IOP > 24 mmHg) on greater than 3 medications.
* Within 1 month prior to screening had YAG laser capsulotomy in the study eye
* Have received any other systemic experimental drug within 12 weeks prior to enrollment.
* Rubeosis iridis or neovascular glaucoma
* Any untreated rhegmatogenous retinal detachment.
* A visual acuity of worse than 20/400 in the fellow eye.
* Unwilling or unable to follow or comply with all study related procedures.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2006-08

PRIMARY OUTCOMES:
To determine the safety and tolerability of 0.5 mg dose of Ranibizumab in the treatment of chronic central serous retinopathy (CSC)

SECONDARY OUTCOMES:
Mean change in VA compared to baseline at month 6 and month 12
Proportion of patients with 20/20 vision at month 6 and 12 as compared to baseline
Proportion of patients losing ≤ 15 letters as measured by ETDRS visual refraction at 4 meters compared to baseline at month 6 and 12
Proportion of patients gaining ≥ 15 letters as measured by ETDRS visual refraction at 4 meters compared to baseline at month 6 and 12
Change in subretinal fluid (as measured by optical coherence tomography) from baseline at month 3, 6, 9 and 12

CONTACTS AND LOCATIONS:
Overall Officials: Richard F. Spaide, M.D., Principal Investigator — Vitreous Retina Macula Consultants of New York, P.C.
Locations (1):
- Vitreous Retina Macula Consultants of New York, P.C., New York, New York, United States